CLINICAL TRIAL: NCT04580823
Title: Exogenous Ketone Salt on Heart and Kidney Ketone Metabolism Measured by Positron Emission Tomography
Brief Title: Heart and Kidney Ketones Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-3441
Record Dates: First submitted 2020-07-07; First posted 2020-10-08 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — Postprandial Period

STUDY DESIGN:
Intervention Model Description: Each participant will have to do the 3 acute interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Fasting without exogenous ketone salt supplement
- Fasting with exogenous ketone salt supplement (Experimental): Fasting with exogenous ketone salt supplement
  Interventions: Dietary Supplement: Fasting with exogenous ketone salt supplement
- Post-Prandial with exogenous ketone salt supplement (Experimental): Post-Prandial with exogenous ketone salt supplement
  Interventions: Dietary Supplement: Post-Prandial with exogenous ketone salt supplement

INTERVENTIONS:
Dietary Supplement: Fasting with exogenous ketone salt supplement — Participants will have to take 2 doses of supplement, one 75 minutes before the scan and one 30 minutes before the scan.
  Other Names: Post-Prandial with exogenous ketone salt supplement
  Arms: Fasting with exogenous ketone salt supplement
Dietary Supplement: Post-Prandial with exogenous ketone salt supplement — Participants will have to take 2 doses of supplement, one 75 minutes before the scan and one 30 minutes before the scan and they will have a liquid meal 20 minutes before the scan.
  Arms: Post-Prandial with exogenous ketone salt supplement

SUMMARY:
Participants will undergo 3 Positron Emission Tomography (PET) scans in 3 different conditions :

1. Fasting without exogenous ketone salt
2. Fasting with exogenous ketone salt supplement
3. Post-Prandial with exogenous ketone salt supplement.

DETAILED DESCRIPTION:
This study will help to quantify heart and kidney ketone uptake with or without an exogenous ketone salt with or without food intake in middle-aged adults. Participants will have 3 different PET scan to perform :

1. Fasting without exogenous ketone salt
2. Fasting with exogenous ketone salt supplement
3. Post-Prandial with exogenous ketone salt supplement.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 45 and 64
* Generally Healthy
* BMI between 18.5 and 27

Exclusion Criteria:

* All drugs taken on a daily basis
* Diabetes or pre-diabetes
* Digestive dysfunction
* Pregnancy or lactation
* Allergy to the supplement
* Participate in an intensive physical exercise training (more than three times a week)
* Being on a ketogenic diet or consumption of ketogenic supplement.
* More than 2 alcoholic beverages each day
* Any clinically significant anomaly in the blood profile
* Smoking
* Claustrophobia
* Being enrolled in another interventional research project or in a PET research project
* Unable to lie dorsally supine for at least 60 minutes

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
11C-Acetoacetate Heart Ketone uptake | 60 minutes
  Heart ketone uptake measured by PET scan
11C-Acetoacetate Kidney ketone uptake | 60 minutes
  Kidney ketone uptake measured by PET scan
Cardiac Functions, telediastolic volume | 60 minutes
  telediastolic volume
Cardiac Functions, telesystolic volume | 60 minutes
  telesystolic volume
Cardiac functions, ejection fraction | 60minutes
  Ejection fraction

SECONDARY OUTCOMES:
Plasma ketone | 60 minutes
  Plasma ketone concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Rearsh Centre on Aging, Sherbrooke, Quebec, Canada